CLINICAL TRIAL: NCT02125279
Title: A Multicenter Open Label Uncontrolled Study of the Long Term Safety and Efficacy of Calcitriol 3 mcg/g Ointment Applied Twice Daily for 26 Weeks in Pediatric Subjects (2 to 16 Years and 11 mo of Age) With Mild to Moderate Plaque Psoriasis
Brief Title: Long Term Safety and Efficacy Study of Calcitriol 3 mcg/g Ointment in Pediatric Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.18131
Record Dates: First submitted 2014-03-28; First posted 2014-04-29 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2019-12

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Calcitriol ointment (Experimental)
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Calcitriol

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of up to 26 weeks of treatment with calcitriol 3 mcg/g ointment when used twice daily, without occlusion, to treat pediatric subjects (2 to 16 years and 11 months of age) with mild to moderate plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 2 to 16 years and 11 months of age
* Clinical diagnosis of stable mild to moderate plaque psoriasis

Exclusion Criteria:

* Other forms of psoriasis
* Hypercalcemia
* Past history of kidney stones
* Vitamin D deficiency
* Other concomitant dermatological disease

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D, LLC
Locations (16):
- United States (8):
  - Johnson Dermatology, Fort Smith, Arkansas
  - Northwest Arkansas Clinical Trials Center, PLLC, Rogers, Arkansas
  - Advanced Skincare Surgery & Medcenter, Burbank, California
  - University of South Florida, Tampa, Florida
  - Shideler Clinical Research Center, Carmel, Indiana
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Montefiore Medical Center, New York, New York
  - Arlington Research Center for Dermatology, Arlington, Texas
- UZ Gent Dermatology Department, Ghent, Belgium
- Canada (2):
  - Lynderm Research Inc., Markham, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
- Germany (3):
  - Charité Universitätsmedizin Berlin, Berlin
  - University Hospital Carl Gustav Carus, Dresden
  - Universitäts-Hautklinik Mainz, Johannes Gutenberg-Universität Mainz, Mainz
- Italy (2):
  - Padova University Hospital, Padua
  - University of Parma, Parma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 88 participants were screened. Only 54 participants out of 88 were enrolled and received study drug, of which 41 participants completed the study.
Groups:
- Calcitriol 3 mcg/g: Participants received calcitriol 3 microgram per gram (mcg/g) ointment applied twice daily without exceeding a maximum of 0.5 gram per kilogram (g/kg) of body weight or 28 gram (g) daily (whichever was the lower) up to 26 weeks. Participants were further followed up for 4 weeks.
Period: Overall Study
Arm/Group | Calcitriol 3 mcg/g
Started | 54
Completed | 41
Not Completed | 13
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Groups:
- Calcitriol 3 mcg/g: Participants received calcitriol 3 mcg/g ointment applied twice daily without exceeding a maximum of 0.5 g/kg of body weight or 28 g daily (whichever was the lower) up to 26 weeks. Participants were further followed up for 4 weeks.
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.3 (3.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 46
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: Participants]
  Canada | 11
  Belgium | 2
  United States | 32
  Italy | 5
  Germany | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Screening in Serum Albumin Levels at Week 4
Description: Change from screening (the last test prior to the first study medication application) in serum albumin levels at week 4 were reported.
Time Frame: Screening, Week 4
Population: Safety population included as all the participants who have applied the study drug at least once. Here 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 48
gram per liter (g/L) | -1.0 (2.28)

2. Primary Outcome: Change From Screening in Serum Albumin Levels at Week 8
Description: Change from screening (the last test prior to the first study medication application) in serum albumin levels at week 8 were reported.
Time Frame: Screening, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 30
g/L | -1.0 (2.09)

3. Primary Outcome: Change From Screening in Serum Albumin Levels at Week 12
Description: Change from screening (the last test prior to the first study medication application) in serum albumin levels at week 12 were reported.
Time Frame: Screening, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 48
g/L | -0.8 (2.03)

4. Primary Outcome: Change From Screening in Serum Albumin Levels at Week 20
Description: Change from screening (the last test prior to the first study medication application) in serum albumin levels at week 20 were reported.
Time Frame: Screening, Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 28
g/L | -1.1 (2.10)

5. Primary Outcome: Change From Screening in Serum Albumin Levels at Week 26
Description: Change from screening (the last test prior to the first study medication application) in serum albumin levels at week 26 were reported.
Time Frame: Screening, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 40
g/L | -0.8 (2.09)

6. Primary Outcome: Change From Screening in Serum Albumin Levels at Week 30 (Follow-up)
Description: Change from screening (the last test prior to the first study medication application) in serum albumin levels at week 30 were reported.
Time Frame: Screening, Week 30 (Follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 16
g/L | -0.2 (2.95)

7. Primary Outcome: Change From Screening in Urine Calcium/Creatinine Ratio at Week 12
Description: Change from screening (the last test prior to the first study medication application) in urine calcium/creatinine ratio at week 12 were reported.
Time Frame: Screening, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 48
Ratio | -0.0164 (0.14340)

8. Primary Outcome: Change From Screening in Urine Calcium/Creatinine Ratio at Week 26
Description: Change from screening (the last test prior to the first study medication application) in urine calcium/creatinine ratio at week 26 were reported.
Time Frame: Screening, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 38
Ratio | 0.0456 (0.15588)

9. Primary Outcome: Change From Screening in Urine Calcium/Creatinine Ratio at Week 30 (Follow-up)
Description: Change from screening (the last test prior to the first study medication application) in urine calcium/creatinine ratio at week 30 were reported.
Time Frame: Screening, Week 30 (Follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 12
Ratio | 0.0715 (0.14333)

10. Primary Outcome: Change From Screening in Serum Phosphate Levels at Week 4
Description: Change from screening (the last test prior to the first study medication application) in serum phosphate levels at week 4 were reported.
Time Frame: Screening, Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 48
mmol/L | 0.0334 (0.17093)

11. Primary Outcome: Change From Screening in Serum Phosphate Levels at Week 12
Description: Change from screening (the last test prior to the first study medication application) in serum phosphate levels at week 12 were reported.
Time Frame: Screening, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 48
mmol/L | 0.0237 (0.17996)

12. Primary Outcome: Change From Screening in Serum Phosphate Levels at Week 20
Description: Change from screening (the last test prior to the first study medication application) in serum phosphate levels at week 20 were reported.
Time Frame: Screening, Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Calcitriol 3 mcg/g: Participants received calcitriol 3 mcg/g ointment twice daily without exceeding a maximum of 0.5 g/kg of body weight or 28 g daily (whichever was the lower) up to 26 weeks.Participants were further followed up for 4 weeks.
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 28
mmol/L | 0.0079 (0.19925)

13. Primary Outcome: Change From Screening in Serum Phosphate Levels at Week 26
Description: Change from screening (the last test prior to the first study medication application) in serum phosphate levels at week 26 were reported.
Time Frame: Screening, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 40
mmol/L | 0.0091 (0.21262)

14. Primary Outcome: Change From Screening in Serum Phosphate Levels at Week 30 (Follow-up)
Description: Change from screening (the last test prior to the first study medication application) in serum phosphate levels at week 30 were reported.
Time Frame: Screening, Week 30 (Follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Calcitriol 3 mcg/g: Participants received calcitriol 3 mcg/g ointment twice daily without exceeding a maximum of 0.5 g/kg of body weight or 28 g daily (whichever was the lower) up to 26 weeks. Participants were further followed up for 4 weeks.
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 16
mmol/L | 0.0145 (0.18727)

15. Primary Outcome: Change From Screening in Serum Parathyroid Hormone (PTH) Levels at Week 4
Description: Change from screening (the last test prior to the first study medication application) in serum PTH levels at week 4 were reported.
Time Frame: Screening, Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Picomole per liter (pmol/L)
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 44
Picomole per liter (pmol/L) | 0.14 (0.967)

16. Primary Outcome: Change From Screening in Serum Parathyroid Hormone Levels at Week 8
Description: Change from screening (the last test prior to the first study medication application) in serum PTH levels at week 8 were reported.
Time Frame: Screening, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 31
pmol/L | 0.09 (1.451)

17. Primary Outcome: Change From Screening in Serum Parathyroid Hormone Levels at Week 12
Description: Change from screening (the last test prior to the first study medication application) in serum PTH levels at week 12 were reported.
Time Frame: Screening, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 48
pmol/L | 0.04 (1.400)

18. Primary Outcome: Change From Screening in Serum Parathyroid Hormone Levels at Week 20
Description: Change from screening (the last test prior to the first study medication application) in serum PTH levels at week 20 were reported.
Time Frame: Screening, Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 28
pmol/L | 0.17 (1.152)

19. Primary Outcome: Change From Screening in Serum Parathyroid Hormone Levels at Week 26
Description: Change from screening (the last test prior to the first study medication application) in serum PTH levels at week 26 were reported.
Time Frame: Screening, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 40
pmol/L | -0.07 (1.744)

20. Primary Outcome: Change From Screening in Serum Parathyroid Hormone Levels at Week 30 (Follow-up)
Description: Change from screening (the last test prior to the first study medication application) in serum PTH levels at week 30 were reported.
Time Frame: Screening, Week 30 (Follow-up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 18
pmol/L | 0.37 (1.796)

21. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is defined as an AE with an onset date on or after the first application of the study drug.
Time Frame: Up to Week 30
Population: Safety population included as all the participants who have applied the study drug at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 54
Participants | 20

22. Secondary Outcome: Number of Participants With Investigator's Global Assessment of Disease Severity (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Each Visit
Description: The IGA is a 0 to 4 point scale. Where, 0 = clear (no signs of psoriasis except for residual hypopigmentation/hyperpigmentation); 1 = almost clear (just perceptible erythema, no induration, and no scaling); 2 = mild (mild erythema, no induration, and mild or no scaling); 3 = moderate (moderate erythema, mild induration, and mild or no scaling); 4 = severe (severe erythema, moderate to severe induration, and scaling of any degree).
Time Frame: Weeks 4, 8, 12, 20, 26 and 30 (Follow-up)
Population: Safety population included as all the participants who have applied the study drug at least once. Here 'N' (overall number of participants analyzed) signifies number of participants evaluable this outcome measure and 'n' (number of participants analyzed) signifies number of participants evaluable for each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 51
Participants
  Week 4 | 3
  Week 8: number analyzed (Participants) | 32
  Week 8 | 5
  Week 12: number analyzed (Participants) | 49
  Week 12 | 15
  Week 20: number analyzed (Participants) | 29
  Week 20 | 14
  Week 26: number analyzed (Participants) | 41
  Week 26 | 19
  Week 30: number analyzed (Participants) | 41
  Week 30 | 17

23. Secondary Outcome: Change From Baseline in Pruritus Score at Each Visit
Description: Pruritus was scored on a 0 to 4 point scale. Where, 0 = none (no-itching); 1 = mild (slight itching, not really bothersome); 2 = moderate (definite itching that is somewhat bothersome without loss of sleep); 3 = severe (intense itching that has caused pronounced discomfort, night rest interrupted); 4 = very severe (very severe itching that has caused pronounced discomfort during the night and daily activities). Positive change from baseline indicate worsening of indication.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 26 and 30 (Follow-up)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 51
Units on a scale
  Week 4 | -0.6 (0.85)
  Week 8: number analyzed (Participants) | 32
  Week 8 | -0.7 (0.64)
  Week 12: number analyzed (Participants) | 49
  Week 12 | -0.7 (0.88)
  Week 20: number analyzed (Participants) | 29
  Week 20 | -0.7 (0.96)
  Week 26: number analyzed (Participants) | 41
  Week 26 | -0.9 (0.98)
  Week 30: number analyzed (Participants) | 41
  Week 30 | -0.8 (1.05)

24. Secondary Outcome: Change From Baseline in Percent (%) Body Surface Area (BSA) at Each Visit
Description: Percent BSA was calculated by modified rules of nines (pediatric participants). Estimate were made from the following for a child up to the age of one year: head and neck total for front and back - 18%; thorax and abdomen-front -18%; thorax and abdomen-back - 18%; each upper limb total for front and back - 9%; each lower limb total for front and back - 14%. For over the age of one year, the relative percentage of BSA changes as follows: the head decreases by 1% per year and the lower limbs increase by 0.5% per year. By the age of ten years, the relative proportions assume the values for adult BSA as follows: perineum becomes 1%; each lower limb becomes a total of 18% front and back; head and neck become 9% total for front and back.
Time Frame: Baseline, Weeks 4, 8, 12, 20, 26 and 30 (Follow-up)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percent BSA
Arm/Group | Calcitriol 3 mcg/g
Number analyzed (Participants) | 51
Percent BSA
  Week 4 | -1.3 (2.85)
  Week 8: number analyzed (Participants) | 32
  Week 8 | -2.5 (4.03)
  Week 12: number analyzed (Participants) | 49
  Week 12 | -3.4 (4.11)
  Week 20: number analyzed (Participants) | 29
  Week 20 | -4.4 (4.61)
  Week 26: number analyzed (Participants) | 41
  Week 26 | -3.9 (4.52)
  Week 30: number analyzed (Participants) | 41
  Week 30 | -4.7 (5.91)

ADVERSE EVENTS:
Time Frame: From start of treatment up to follow up (30 weeks)
Arm/Group | Calcitriol 3 mcg/g
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 9/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Calcitriol 3 mcg/g (N=54)
Nasopharyngitis (Infections and infestations) | 6
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-01-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT02125279/Prot_000.pdf
  • Statistical Analysis Plan (2014-05-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT02125279/SAP_001.pdf